CLINICAL TRIAL: NCT02528916
Title: Nociceptin Concentration in Synovial Fluid and Plasma in Patients Undergoing Primary Total Knee Arthroplasty: A Prospective Pilot Study
Brief Title: Nociceptin Concentration in Synovial Fluid and Plasma
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Julia Caldwell, Assistant Professor of Anesthesiology, Milton S. Hershey Medical Center
Other Study IDs: 42679
Record Dates: First submitted 2015-07-05; First posted 2015-08-19 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Knee Arthroplasty Patients: Patients who consented, met inclusion and exclusion criteria, had plasma and synovial fluid samples drawn as described in the included protocol. No interventions were completed. No changes to standard of care treatment completed.

SUMMARY:
Nociceptin/Orphanin is a novel opioid peptide system associated with inflammatory response. Currently is it uncertain as to the presence of absence of nociceptin in synovial fluid of patients. Nociceptin levels will be measured pre-operatively and post-operatively in plasma levels of patients receiving primary total knee arthroplasty. Nociceptin levels will also be measured in synovial fluid levels prior to surgical manipulation.

DETAILED DESCRIPTION:
This is a prospective observational study where nociceptin levels will be drawn from the patient's serum as well as from the patient's synovial fluid. The blood draws will be completed by the anesthesia team and the synovial fluid and tissue will be obtained by the orthopedic team. The initial blood draw will be in the preoperative area and the second blood draw will be five minutes after the release of the tourniquet. The synovial fluid will be drawn by the surgeon with the first incision. There will be no randomization nor control group.

Endpoints:

1. The level or absence of nociceptin in synovial fluid in patients receiving total knee primary arthroplasty will be measured via ELISA in picograms per volume.
2. The level or absence of nociceptin in plasma in patients receiving total knee primary arthroplasty both in the preoperative period (less than 1 hour prior to surgery and 5 minutes after the tourniquet is removed) via ELISA in picograms per volume.
3. Determine the changes if any of nociception plasma levels during the perioperative course of patients receiving total primary knee arthroplasty.

Secondary Study Endpoints:

1. Determine the effect if present of history of chronic pain and opioid use on the levels of nociception present in patients' synovial fluid and plasma receiving primary total knee arthroplasty.
2. Determine the effect if present of demographic factors on the levels of nociception present in patients' synovial fluid and plasma receiving primary total knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* receiving a primary knee joint arthroplasty by Dr. Davis ages 18-80 years hemodynamically stable no joint or other types of infection informed consent received and signed no prior joint arthroplasty at the current surgical site no other surgical intervention planned

Exclusion Criteria:

* prior knee arthroplasty at site outside of desired age range pregnant current infection in joint or other location no desire to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sequential patients receiving primary unilateral knee arthroplasty by the same surgeon
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Nociceptin in Synovial Fluid | The surgeon will make a small incision after the patient has been anesthetized and prepped and draped. He will then withdraw the synovial fluid and then will begin the surgery after the fluid is removed.
  The level or absence of nociceptin in synovial fluid will be measured using ELISA and represented in picograms per volume.

SECONDARY OUTCOMES:
Nociceptin in Plasma | Blood will be drawn in the preoperative period (approximately up to 1 hour prior to surgery).
  Determine the presence of absence of nociceptin in plasma in patients receiving total knee primary arthroplasty and determine the changes if any of nociception plasma levels during the perioperative course of patients receiving total primary knee arthroplasty. Nociceptin will be measured using ELISA and represented in terms of picograms per volume.
Nociceptin in Plasma | Blood will be drawn 5 minutes after the release of the tourniquet.
  Determine the presence of absence of nociceptin in plasma in patients receiving total knee primary arthroplasty and determine the changes if any of nociception plasma levels during the perioperative course of patients receiving total primary knee arthroplasty. Nociceptin will be measured using ELISA and represented in terms of picograms per volume.
Patient Demographics | Will be determined in the preoperative period up to one hour prior to surgery.
  Age
Patient Demographics | Will be determined in the preoperative period up to one hour prior to surgery.
  Gender
Patient Demographics | Will be determined in the preoperative period up to one hour prior to surgery
  BMI
Patient Pain Scores | One set of preoperative scores will be obtained up to one hour prior to surgery.
  pre-operative pain scores will be determined using the 0-10 verbal analog scale.
Patient Pain Scores | One set of post operative pain scores will be obtained up to one hour post emergence from anesthesia.
  post-operative pain scores will be determined using the 0-10 verbal analog scale.

REFERENCES:
- [Background] Chiou LC, Liao YY, Fan PC, Kuo PH, Wang CH, Riemer C, Prinssen EP. Nociceptin/orphanin FQ peptide receptors: pharmacology and clinical implications. Curr Drug Targets. 2007 Jan;8(1):117-35. doi: 10.2174/138945007779315605. PMID 17266536
- [Background] Lin AP, Ko MC. The therapeutic potential of nociceptin/orphanin FQ receptor agonists as analgesics without abuse liability. ACS Chem Neurosci. 2013 Feb 20;4(2):214-24. doi: 10.1021/cn300124f. Epub 2012 Nov 6. PMID 23421672
- [Result] Kumar N, Smart D, Mason S, McKnight AT, Rowbotham DJ, Lambert DG. Neither nociceptin nor its receptor are present in human synovial fluid or tissue. Br J Anaesth. 1999 Sep;83(3):470-1. doi: 10.1093/bja/83.3.470. PMID 10655922
- [Derived] Verbeek TA, Jarbadan NR, Davis C, Caldwell J. Nociceptin is present in synovial fluid of patients undergoing total knee arthroplasty. J Orthop Surg Res. 2020 Jul 16;15(1):266. doi: 10.1186/s13018-020-01789-1. PMID 32677997